CLINICAL TRIAL: NCT00858377
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered AMG 900 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 First-in-Human Study Evaluating AMG 900 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080016
Record Dates: First submitted 2009-02-26; First posted 2009-03-09 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Solid Tumors; Tumors
Keywords: Amgen; Phase 1; First in Human; Advanced Solid Tumors; Clinical Trial; Aurora kinase inhibitor; Open-label; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1- Dose Expansion (Experimental): The dose expansion part of the study will begin after completion of the dose escalation phase and will consist of 3 cohorts of 14 subjects each. One taxane-resistant tumor type will be evaluated in each cohort.
  Interventions: Drug: Arm 1- Dose Expansion
- Arm 1- Dose Escalation (Experimental): The dose escalation part of the study is aimed at determining the maximum tolerated dose (MTD) of AMG 900 and if necessary, the MTD with prophylactic GCSF support (MTD-G).
  Interventions: Drug: Arm 1- Dose Escalation

INTERVENTIONS:
Drug: Arm 1- Dose Escalation — AMG 900 is a small molecule inhibitor of aurora kinases A, B and C. AMG 900 will be administered daily for 4 days every 2 weeks (i.e., 4 consecutive days of dosing followed by 10 consecutive days off treatment).
  Arms: Arm 1- Dose Escalation
Drug: Arm 1- Dose Expansion — AMG 900 is a small molecule inhibitor of aurora kinases A, B and C. AMG 900 will be administered daily for 4 days every 2 weeks (i.e., 4 consecutive days of dosing followed by 10 consecutive days off treatment).
  Arms: Arm 1- Dose Expansion

SUMMARY:
This first-in-human study of AMG 900 will be conducted in two parts: dose escalation and dose expansion. The dose escalation part of the study is aimed at evaluating the safety, tolerability and PK of oral AMG 900 in subjects with advanced solid tumors. Up to 50 subjects may be enrolled in dose escalation. The dose expansion part of the study will consist of 42 subjects in three taxane-resistant tumor types. The dose of AMG 900 will be dependent upon data from the dose escalation part of the study

DETAILED DESCRIPTION:
that G-CSF must be started at day 5, 1 day after the last day of AMG 900 and be continued until neutrophiles are > 1000 or until day 12, meaning 2 days before the reinduction.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Part 1 Dose Escalation only: advanced solid tumor refractory to standard treatment for which no standard therapy is available or the subject refuses standard therapy
* Part 1 Dose Escalation only: Measurable or evaluable disease per RECIST guidelines
* Part 2 Dose Expansion only: Taxane-resistant tumor (defined as refractory to or progression within 6 months of discontinuing paclitaxel or docetaxel) of prespecified histology
* Part 2 Dose Expansion only: Measurable disease per RECIST guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Life expectancy of > 3 months, in the opinion of the investigator
* Willing to provide existing and/or future paraffin-embedded tumor samples
* Part 1 Dose Escalation: must have tumor tissue that is accessible for biopsy by fine needle aspiration (FNA) and must consent to undergo biopsies of their tumor (subjects in non-accelerated phase only)
* Ability to take oral medications
* Competent to sign and date an Institutional Review Board approved informed consent form
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Hemoglobin > 9 g/dL
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN)
* Serum creatinine < 2.0 mg/dL
* Calculated creatinine clearance ≥ 50 ml/min
* AST < 2.5 x ULN (if liver or bone metastases are present, ≤ 5 x ULN)
* ALT < 2.5 x ULN (if liver or bone metastases are present, ≤ 5 x ULN)
* Alkaline phosphatase < 2.0 x ULN (if liver or bone metastases are present, ≤ 5 x ULN)
* Total bilirubin < 1.5 x ULN

Exclusion Criteria:

* Active parenchymal brain metastases. Subjects who have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to study day 1 are eligible if they meet all of the following criteria: a) residual neurological symptoms grade < 1; b) no dexamethasone requirement; and c) follow-up MRI shows no new lesions appearing
* Prior bone marrow transplant (autologous or allogeneic)
* History or presence of hematological malignancies
* History of bleeding diathesis
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Active peptic ulcer disease
* Gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (eg, Crohn's disease, ulcerative colitis)
* Active infection requiring intravenous (IV) antibiotics within 2 weeks of study enrollment (day 1)
* Known positive test for HIV
* Active or chronic hepatitis B or hepatitis C infection, determined by serologic tests
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia
* Anti-tumor therapy within 28 days of study day 1; concurrent use of hormone deprivation therapy for hormone-refractory prostate cancer or breast cancer is permitted
* Treatment with immune modulators including, but not limited to, corticosteroids, cyclosporine and tacrolimus within two weeks prior to enrollment
* Therapeutic or palliative radiation therapy within two weeks of study day 1
* Systemic anticoagulation therapy, including warfarin, within 28 days of day 1
* Prior treatment with aurora inhibitors
* Prior participation in an investigational study (drug or device) within 28 days of study day 1
* Major surgery within 28 days of study day 1
* Any co-morbid medical disorder that may increase the risk of toxicity, in the opinion of the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-08-10 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Safety: subject incidence of adverse events, first-cycle DLTs and clinically significant changes in vital signs, weight, ECGs and clinical laboratory tests | 1 year
PK profile: AMG 900 PK parameters including, but not limited to, maximum observed concentration (Cmax), minimum observed concentration, area under the plasma concentration-time curve and, if feasible, half-life | 1 year
Change in levels of p-Histone H3 from baseline (part 1 - dose escalation only) | 1 year
Response rate in each taxane-resistant tumor type assessed per RECIST guidelines (part 2 - dose expansion only) | 1 year

SECONDARY OUTCOMES:
Change in tumor volume from baseline measured by volumetric CT or MRI | 1 year
Tumor response measured by CT or MRI and assessed per RECIST guidelines | 1 year
Change from baseline in maximum standardized uptake value (SUVmax) using 18FLT-PET/CT (part 2 - dose expansion only) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (5):
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Baltimore, Maryland
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
- Australia (3):
  - Research Site, Kurralta Park, South Australia
  - Research Site, Bentleigh East, Victoria
  - Research Site, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Carducci M, Shaheen M, Markman B, Hurvitz S, Mahadevan D, Kotasek D, Goodman OB Jr, Rasmussen E, Chow V, Juan G, Friberg GR, Gamelin E, Vogl FD, Desai J. A phase 1, first-in-human study of AMG 900, an orally administered pan-Aurora kinase inhibitor, in adult patients with advanced solid tumors. Invest New Drugs. 2018 Dec;36(6):1060-1071. doi: 10.1007/s10637-018-0625-6. Epub 2018 Jul 7. PMID 29980894
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com